CLINICAL TRIAL: NCT03608176
Title: Evaluation of the Efficacy of Plant-based Approaches to Stop Obesity Diet in Comparison With a Control Group on Body Weight in Mexican Adults With Overweight and Obesity: Randomized Controlled Trial
Brief Title: Evaluation of the Plant-based Approaches to Stop Obesity Diet for the Treatment of Overweight and Obesity
Acronym: PASO diet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Sonora (Other)
Responsible Party: Principal Investigator, Rolando Giovanni Díaz Zavala, Principal Investigator, Universidad de Sonora
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PASOdiet-OBMEX-2018
Record Dates: First submitted 2018-07-23; First posted 2018-07-31 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Overweight and Obesity
Keywords: Obesity; Randomized Controlled Trial; Lifestyle Intervention; Plants; Water; Weight loss; Diet; Overweight
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PASO diet group (Experimental)
  Interventions: Other: PASO diet group
- Low-fat diet group (Active Comparator)
  Interventions: Other: Low-fat diet group
- Waiting list group (Other)
  Interventions: Other: Waiting list group

INTERVENTIONS:
Other: PASO diet group — This group include a low-fat, low calorie diet (1200-1800 kcal), in addition of a behavioral change protocol. They will also be instructed to consume green tea (2 cups/day for 3 days/week), black tea (2 cups/day for 2 days/week), coffee (2 cups/day for 2 days/week), cinnamon (1 tsp/day for at least 3 days/week), psyllium fiber (3 tsp/day/week) and water (1.5 L/day/week).
  Arms: PASO diet group
Other: Low-fat diet group — This group include a low-fat, low calorie diet (1200-1800 kcal), in addition of a behavioral change protocol.
  Arms: Low-fat diet group
Other: Waiting list group — This group will only receive written information with recommendations on healthy eating. When the study finished, this group will receive a behavioral change protocol with a low-fat, low calorie diet.
  Arms: Waiting list group

SUMMARY:
The accumulation of excess of body weight is one of the most important problems worldwide, thus effective and accessible treatments are required. Some authors highlighted that treatment is focused solely on lifestyle (diet, physical activity, behavioral therapy) has a limited effect on body weight because it does not consider the biological mechanisms linked to weight loss in patients with obesity. On the other hand, drugs and bariatric surgery consider these biological approaches; however, its costs, safety and effectiveness limits its use on a large scale. Research studies support the existence of compounds in plants (such as epigallocatechin gallate, caffeine, cinnamaldehyde, fiber), and water with biological properties that would contribute to the treatment of overweight and obesity. However, at the moment, these compounds have only been evaluated individually and their effects have been significant but limited clinically, therefore, more research studies are needed to evaluate whether several of these compounds contained in common plants synergistically have a clinical impact on the management of overweight and obesity. The present work integrates diverse plant-based approaches to stop obesity and it is compared with a control group and a waiting list group. The main aim is to evaluate the efficacy of the Plant-based Approaches to Stop Obesity diet (PASO diet) compared with a control group on body weight at 3 months in Mexican adults with overweight and obesity. This is a pilot study designed as a randomized controlled trial. The study will be conducted with a (n=36). The primary outcome is the change in body weight from baseline to 3 months. Secondary outcomes will be the changes from baseline to 3 months in body mass index, waist circumference, systolic and diastolic blood pressure, symptoms of depression, quality of life scales and biochemical parameters (fasting glucose, total cholesterol, LDL cholesterol, HDL-cholesterol, triglycerides and gamma glutamyl transferase). Additionally two 24-hour dietary recall will be measured at baseline and 3 months to evaluate adherence to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Mexican adults (> 20 years and <55)
* Residents of the city of Hermosillo, Sonora
* Obesity (BMI> 25 and <45)
* Availability of time to participate in the study.
* Economic capacity to acquire the assigned diet
* Grant informed consent
* Keep a dietary record for one week prior to the intervention

Exclusion Criteria:

* Medical conditions that constitute a contraindication for the intervention, such as de-controlled diabetes, dyslipidemia with pharmacological treatment, blood pressure ≥160 / 100 mmHg, heart failure, renal failure, etc.
* Previous bariatric surgery
* Participate in another intervention or treatment for the management of obesity
* Use of drugs or substances with an effect on weight, for example, metformin, orlistat or corticoids
* Weight loss> 5% of total body weight in the last 4 months
* Pregnancy or lactation
* Another member of the family or acquaintance who has agreed to participate in the study
* Consumption of more than 10 alcoholic drinks per week
* Use of addictive substances as drugs of abuse
* Psychiatric condition that prevents adherence to treatment, such as severe depression, bipolarity and schizophrenia Illiteracy
* Gastrointestinal problems or any condition where coffee, tea or cinnamon are not well tolerated or contraindicated
* People who drink more than 4 cups of coffee (tea) per day or its equivalent in caffeinated beverages.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in body weight | baseline to 3 months

SECONDARY OUTCOMES:
Change in waist circumference | baseline to 3 months
Change in body fat percentage | baseline to 3 months
Change in the Beck Depression Inventory score | baseline to 3 months
  The Beck Depression Inventory (BDI) is a 21-item questionnaire that assesses mood over the previous week. Total scores range from 0 to 63, with higher values indicating greater symptoms of depression. Scores of 0-9 reflect minimal (subclinical) symptoms, values of 10-18, 19-29, and ≥30 indicate mild, moderate, and severe symptoms of depression, respectively.
Change in the Short Form-36 Health Survey score | baseline to 3 months
  The SF-36 Health Survey evaluates aspects of the quality of life in adult populations (over 16 years of age). The result of its application is the generation of eight concepts or scales of health, result of the average of the sum of the questions contained in the questionnaire for each concept. These concepts are: physical function, physical role, corporal pain, general health, vitality, social function, emotional role and mental health. The SF-36 is a self-applied instrument and contains 36 questions. For each scale, the answers to each question are coded and recoded (10 questions), and the results are interpreted on a scale of 0 to 100, lower results indicate poorer health and greater result better health).
Change in systolic and diastolic blood pressure | baseline to 3 months
Change in fasting glucose | baseline to 3 months
Change in total cholesterol | baseline to 3 months
Change in LDL-cholesterol | baseline to 3 months
Change in HDL-cholesterol | baseline to 3 months
Change in triglycerides | baseline to 3 months
Change in gamma glutamyl transferase | baseline to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Rolando G Díaz Zavala, Ph.D., Principal Investigator — Universidad de Sonora
Locations (1):
- Centro de Promoción de Salud Nutricional (CPSN), Hermosillo, Sonora, Mexico

IPD SHARING:
Plan to Share IPD: Undecided